CLINICAL TRIAL: NCT03908840
Title: An Open-label, Multicenter, Phase 1 Study of TBI 302 as Second-Line Therapy in Patients With Non-resectable, Non-transplantable, Non-radiofrequency Ablation (RFA) Treatable Hepatocellular Carcinoma (HCC)
Brief Title: Open-label Multicenter Phase 1 Study of TBI 302 as Second-Line Therapy in Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Therapure Biopharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBI 302-001
Record Dates: First submitted 2012-08-17; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular; Carcinoma; Liver; Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TBI 302 Safety, Tolerability (Experimental): 5 Cohorts, Dose escalation TBI 302 will be formulated in 0.9% saline. TBI 302 in a syringe will be administered over approximately 1 hour under constant observation once per week for 4 weeks (on Days 1, 8, 15 and 22).
  Interventions: Biological: TBI 302

INTERVENTIONS:
Biological: TBI 302 — TBI 302 administered once a week in first 3 weeks and no treatment in week 4 (28 days is 1 cycle). Followed once weekly treatment of TBI 302 for 3 weeks followed by no treatment in week 4 (cycle 2)

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common cancers worldwide. TBI 302 is being developed for the treatment of inoperable HCC by intravenous infusion. The objective is to determine the safety and tolerability of TBI 3002.

DETAILED DESCRIPTION:
This is an open-label, Phase 1 study to evaluate the safety, tolerability, PK, and MTD of TBI 302 in patients with non-resectable, non-transplantable HCC. Tumor response will be assessed at Week 9 (5 weeks following cessation of treatment) according to RECIST (ver 1.1) and AASLD criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients histologically or cytologically confirmed, unresectable, or metastatic HCC
* Child-Pugh Category A or B (score 6-7); stable, well-compensated, mild cirrhosis with minimal or no ascites
* Male or female patients 18 years of age or older
* Patients must be willing and able to read, understand and sign a written informed consent form
* Male, or female of childbearing potential, must agree to use double barrier contraception, oral contraceptives or other ways to avoid pregnancy during the study and for 90 days after the last day of treatment
* Life expectancy of greater than 3 months
* Plasma haptoglobin ≥ LLN (lower limit of normal)

Exclusion Criteria:

* Patients confirmed with hemolysis confirmed by serum lactate dehydrogenase, serum haptoglobin or indirect bilirubin levels
* Patients who have received a blood transfusion within 4 weeks of enrolment
* Patients with infiltrating diffuse hepatocellular carcinoma, Type 1 or 2 diabetes mellitus, Hepatitis B or Hepatitis C infection
* Systemic chemotherapy-naive patients
* Patients with significant cardiovascular impairment, including history of congestive heart failure, unstable angina, myocardial infarction, or serious cardiac arrhythmia within the last 6 months
* Patient with a history of tumor rupture
* Patients with serious non-healing wound , ulcer or bone fracture
* Known positive human immunodeficiency virus (HIV) test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) observed during the trial | through study completion, up to one year
  The number of TEAEs observed during the trial

SECONDARY OUTCOMES:
Determination of Maximum Tolerated Dose | through study completion, up to one year
  Determination of Maximum Tolerated Dose of TBI 302

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States